CLINICAL TRIAL: NCT02325921
Title: Advanced MRI in Renal Tumors.
Brief Title: MRI in Renal Tumors
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL49616.091.14
Record Dates: First submitted 2014-12-02; First posted 2014-12-25 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Magnetic Resonance Imaging; Diffusion Weighted MRI; Diffusion Tensor Imaging
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal tumor.: Patients >18 years of age with histopathologically confirmed renal tumor diagnosis.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — One MRI examination, diagnostic scanning protocol as used for renal tumours with additional diffusion weighted sequences, but without contrast enhancement.

SUMMARY:
Diagnostic imaging for renal masses of unknown nature using conventional imaging modalities such as 3 phase contrast-enhanced computed tomography (CT) is not always conclusive. After (partial) nephrectomy, 10-20 % of the resected tumors show benign histology which could not be identified on diagnostic imaging. With improved imaging techniques available, leading to improvements in characterisation of renal tumors, the number of unnecessary resections may be reduced. The objective of this study is to assess the ability to discriminate oncocytoma from RCC based on the ADC distribution parameters with addition of, tumor volume, and patient demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic diagnosis of renal tumor based on previous ultrasonography, CT or MRI examinations.
* Signed Institutional Review Board (IRB) approved informed consent form.
* Being at least 18 years of age.
* Histopathologically confirmed renal tumor diagnosis.

Exclusion Criteria:

* Relative contra indications for MRI (metal device/foreign bodies, claustrophobia);
* Active renal or perirenal infection;
* Minor and/or incapacitated adult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients >18 years of with a histopathologically confirmed renal tumor diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Discriminating malignant from benign renal lesions using Apparent Diffusion Coefficient (ADC, a metric obtained by diffusion weighted MRI) value distribution analysis. | 45 months

SECONDARY OUTCOMES:
Additional value of tumor volume and patient characteristics to discriminate malignant from benign renal lesions. | 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen J. Futterer, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands